CLINICAL TRIAL: NCT06650540
Title: Levofloxacin Plus Metronidazole Suppositories Versus Levofloxacin Co-administered with Metronidazole Tablets for the Treatment of Chronic Endometritis: a Randomized Controlled Trial
Brief Title: Levofloxacin Plus Metronidazole Suppositories Versus Levofloxacin Co-administered with Metronidazole Tablets in Chronic Endometritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Lin MingMei, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT of chronic endometritis; No. BYSY2023022 (Other Grant/Funding Number: Key Clinical Projects of Peking University Third Hospital)
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: IVF
Keywords: Chronic Endometritis; pregnancy outcomes; pharmacological treatment
MeSH Terms: interventions — Levofloxacin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levofloxacin Plus Metronidazole Suppositories group (Experimental): Clinical pregnancy outcomes of the first embryo transfer in patients with chronic endometritis treated with Levofloxacin Plus Metronidazole Suppositories.
  Interventions: Drug: Levofloxacin Plus Metronidazole Suppositories
- Levofloxacin co-administered with Metronidazole tablets group (Active Comparator): Clinical pregnancy outcomes after the first embryo transfer in patients with chronic endometritis treated with Levofloxacin co-administered with Metronidazole tablets.
  Interventions: Biological: Levofloxacin co-administered with Metronidazole tablets

INTERVENTIONS:
Drug: Levofloxacin Plus Metronidazole Suppositories — Administer a two-week course of Levofloxacin Plus Metronidazole Suppositories to patients diagnosed with chronic endometritis.
  Other Names: Experimental
  Arms: Levofloxacin Plus Metronidazole Suppositories group
Biological: Levofloxacin co-administered with Metronidazole tablets — Administer a two-week course of Levofloxacin in combination with Metronidazole tablets to patients diagnosed with chronic endometritis.
  Other Names: Active Comparator
  Arms: Levofloxacin co-administered with Metronidazole tablets group

SUMMARY:
This is a single randomised controlled trial. The investigators plan to randomise 800 participants to the levofloxacin plus metronidazole suppositories versus levofloxacin co-administered with metronidazole tablets for the treatment of chronic endometritis in a 1:1 rate. Primary outcome will be the live birth rate after the embryo transfer.

DETAILED DESCRIPTION:
Chronic endometritis (CE) is a pathological condition characterized by inflammation and destruction of the endometrium. In this disease state, microorganisms coexist with the host's immune system in a balanced manner. However, for the majority of patients with CE, clinical symptoms are nonspecific and atypical, rendering diagnosis based on clinical signs or blood tests unreliable. Consequently, invasive procedures such as histopathological examination of the endometrium or hysteroscopy are often necessary to establish a definitive diagnosis. The infiltration of plasma cells in the endometrial stroma associated with CE, together with increased production of immunoglobulins and pro-inflammatory cytokines, can reduce endometrial receptivity. This reduction in receptivity can lead to an increased risk of female infertility, lower pregnancy rates, and reduced live birth rates, which are linked to unexplained infertility, repeated failure of embryo implantation, and recurrent miscarriages. While the etiology of CE remains elusive, it is widely believed to be related to infection by pathogenic microorganisms such as Streptococcus, Enterococcus faecalis, Escherichia coli, Staphylococcus , Klebsiella pneumoniae, Ureaplasma, and Mycoplasma, which can ascend from the vagina into the uterine cavity. Preliminary basic research by investigators also supports the notion that bacterial infections are a leading cause of endometritis. The mainstay of CE treatment currently involves oral antibiotics, with a common regimen being colabitux (500 mg once daily for 14 days) in combination with metronidazole (400 mg twice daily for 14 days). However, oral antibiotics can face issues such as drug resistance, suboptimal local concentrations of the drug, and a propensity to cause gastrointestinal side effects like nausea, vomiting, diarrhea, abdominal distension, and dermatological reactions like skin rashes and leukopenia, which can lead to treatment interruptions and reduced efficacy in managing chronic endometritis. Therefore, there is a need to explore methods to enhance the treatment success rate of CE. Metronidazole suppositories, composed primarily of metronidazole, are used vaginally to treat bacterial infections and other types of bacterial-induced vaginitis. Acting directly on the local area, these suppositories typically exhibit faster and more pronounced therapeutic effects without adversely affecting other tissues and organs. Given that the vagina is connected to the uterine cavity via the cervix, investigators hypothesized that local vaginal administration of the medication might be more effective. This approach not only achieves higher local concentrations of the drug in the uterine cavity, but also prevents ascending infection of vaginal bacteria.

In the prospective, randomized study conducted by investigators, the efficacy of levofloxacin plus metronidazole suppository versus levofloxacin co-administered with metronidazole tablets was compared in patients with chronic endometritis. By comparing the pregnancy outcomes of the two groups, the aim was to identify a superior treatment strategy, enhance treatment efficacy, and improve clinical outcomes.

Purpose The objective of this study is to investigate the efficacy of metronidazole therapy in enhancing treatment outcomes for chronic endometritis, with the aim of increasing clinical pregnancy and live birth rates in IVF procedures, reducing miscarriage rates, and thereby offering a safer and more effective treatment option for participants with chronic endometritis who are considering pregnancy.

Design This study is designed as a randomized controlled trial. Study Population

Inclusion Criteria:

1. Infertile participants between the ages of 20 and 42.
2. Participants who have undergone hysteroscopy and endometrial biopsy, resulting in a pathological diagnosis of chronic endometritis.
3. Participants with a blood FSH level of 12 U/L on the second day of their menstrual cycle.
4. Participants who have provided informed consent and signed the consent form.

Exclusion Criteria:

1. Participants diagnosed with uterine submucosal fibroids, a history of uterine malformations or previous corrective surgeries for such deformities, uterine intrauterine adhesions, or a history of pelvic tuberculosis or endometrial tuberculosis, including cases with pathology suggesting endometrial tuberculosis.
2. Participants or their partners with a history of fetal or child chromosomal abnormalities and those planning a pre-implantation genetic screening.
3. Participants with a well-documented clear history of allergy to the study medication.

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients aged 20-42 years
* Hysteroscopy and endometrial biopsy were performed, and the
* Pathological diagnosis was chronic endometritis
* Serum FSH level on the second day of menstruation was ≤12U/L
* Agree and sign the informed consent form

Exclusion Criteria:

* Patients with the following diagnoses: submucosal myoma; Uterine malformation or previous surgery for correction of uterine deformity; Intrauterine adhesions; The previous history of pelvic tuberculosis or endometrial tuberculosis or the current pathology suggested endometrial tuberculosis; Endometrial hyperplasia or endometrial cancer
* Patients with spouse, previous fetal or child chromosomal abnormalities who plan to undergo preimplantation genetic screening
* Patients with a history of allergy to study drugs

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 800 (Estimated)
Dates: Start 2024-10-22 (Estimated); Primary Completion 2025-10-22 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
live birth rate after the first embryo transfer | 22 weeks to 43 weeks gestation after the first embryo transfer cycle
  Live birth is defined as the delivery of at least one baby after 22 weeks of gestation Oversight that exhibits any sign of life.

SECONDARY OUTCOMES:
Clinical pregnancy | around 7 weeks' gestation after the first embryo transfer cycle
  It is defined as at least one gestational sac on ultrasound at around 7 weeks'gestation with the detection of heart-beat activity,
Ongoing pregnancy | 12 weeks to 43weeks gestation after the first embryo transfer cycle
  definedIs pregnancy with detectable heart rate at 12 weeks' gestation or beyond
Biochemical pregnancy | about 14 days after embryo transfer
  defined as a positive pregnancy test
Miscarriage | 6-22 weeks of gestation
  defined as spontaneous loss of a clinical pregnancy before 22 completed weeks of gestational age, in which the embryo(s) or fetus(es) is/are nonviable or is/are absorbed or expelled from the uterus.
Cumulative live birth | 6 monti after the first embryo transfer
  the cumulative rate of live bor children conceived within six months of the first FET cycle.
Pre-eclampsia | after 20 weeks of gestation
  defined as the development of gestational hypertension with proteinuria (≥300 mg/24-hour urine collection or 30 mg/dL. in single urine sample) of new onset after 20 weeks of gestation
Gestational hypertension | after 20 weeks of gestation
  defined as the development of blood pressure greater than 140/90 mmHg after pregnancy without proteinuria or other signs of preeclampsia Time Frame: after 20 weeks of gestation
Gestational diabetes mellitus | between 24 -28 weeks of gestation
  defined as carbohydrate intolerance of variable severity with onset or first recognition during pregnancy as determined from the diagnosis in the obstetrical medical record
Premature rupture of membrane(PROM)rate | Time Frame: the day of delivery
  defined as rupture of the amniotic membranes before the onset of labor including Measures PROM at term and preterm PROM
Preterm delivery | up to 37 weeks
  defined as delivery of a fetus at less than 37 weeks' gestational age
Placenta previa | the day of delivery
  defined as a placenta that is implanted over or very close to the internal cervical orifice
Postpartum hemorrhage | the day of delivery
  defined as the loss of 500 ml of blood or more after completion of the third stage of labor
Birth weight | the day of delivery
  Birth weight
Stillbirth | the day of delivery
  defined > the absence of signs of life at or after birth
Mode of delivery | the day of delivery
  Veginal birth or Caesereen Section

CONTACTS AND LOCATIONS:
Locations (1):
- Peking university third hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Results of the study will be submitted to scientific conferences in reproductive medicine and a peer-reviewed journal.
Supporting Information: Study Protocol, SAP
Time Frame: the day of publishing the main results, Around 3 years from now
Access Criteria: please contact the hukailun@bjmu.edu and linmingmei2023@163.com

REFERENCES:
- [Derived] Lin M, Wang Y, Lv X, Lin Z, Zeng Z, Mo D, Shan H, Li R. Administration of levofloxacin combined with metronidazole suppositories prior to in vitro fertilisation in women with chronic endometritis: a protocol of a single-centre, randomised, controlled clinical trial. BMJ Open. 2025 Sep 15;15(9):e098500. doi: 10.1136/bmjopen-2024-098500. PMID 40954081